CLINICAL TRIAL: NCT01303939
Title: Neuroimaging Brain Changes in Glaucoma
Brief Title: Does Glaucoma Cause Loss of Brain Function?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal Investigator, Wills Eye
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-009
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma
Keywords: Glaucoma; MRI Brain Scan; Voxel-Based Morphometry
MeSH Terms: conditions — Glaucoma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Magnetic resonance images (MRI) of the brain were obtained from glaucoma patients to look at structures and volume. Age, gender, ethnic healthy matches for each glaucoma patient received MRIs of the brain for comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Glaucoma Patients (Other): Patients who were outliers from two previous studies: Assessment of Ability Related to Vision (AARV) or Assessment of Disability Related to Vision (ADREV) with mini mental status exam score of 25 or higher underwent magnetic resonance imaging (MRI) of the brain to look at structures and volume.
  Interventions: Diagnostic Test: magnetic resonance imaging (MRI) of the brain
- Control Patients (Other): Age, gender and race matched (to each glaucoma patient) group of healthy individuals with no ocular diseases with mini mental status exam score of 25 or higher underwent magnetic resonance imaging (MRI) of the brain to look at structures and volume.
  Interventions: Diagnostic Test: magnetic resonance imaging (MRI) of the brain

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging (MRI) of the brain — High resolution three-dimensional T1-weighted magnetic resonance imaging (MRI) was obtained from each participant at one visit.
  Other Names: Brain MRI

SUMMARY:
The purpose of the study is to determine if glaucoma is associated with neurodegenerative changes in areas of the brain other than the occipital lobe. This will help guide the direction of further research in the use of neuroprotective agents in preventing or controlling such changes. The final goal is to improve the quality of life for patients with glaucoma.

DETAILED DESCRIPTION:
Death of retinal ganglion cells causes loss of neurons in areas other than just the visual cortex. These neurodegenerative changes decrease the patient's ability to perform the activities of daily living. Tensor-based morphometry analysis of magnetic resonance imaging (MRI) brain scans will reveal areas of cortical degeneration in glaucoma patients, and the extent of damage in these areas should correlate with patients ability to perform vision-dependent tasks, as measured by the Assessment of Ability Related to Vision (AARV).

Patients with glaucoma who were outliers in two previous studies, Assessment of Ability Related to Vision (AARV) or Assessment of Disability related to vision (ADREV), in that they had poor performance-based measure scores despite having midrange visual field scores.

Mini-Mental State Exam and T-1 weighted MRI brain scan and will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma who were participated in other studies Assessment of Ability Related to Vision (AARV) or Assessment of Disability Related to Vision (ADREV) and were found to be outliers in that they have poor performance-based measure scores (≤ 40) despite having midrange visual field scores (mean deviation of -6 to -20).
* Age-, gender- and race-matched controls who do not have glaucoma, and who do not have loss of vision for any reason other than cataract or refractive error.

Exclusion Criteria:

1. Patients with any type of neurological disease.
2. Patients with a cognitive deficit which would affect visual functioning, as revealed by score of less than 25 in the mini mental status examination.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Glaucoma Service, Wills Eye Institute
Locations (1):
- Wills Eye Institute, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lackey J, Williams AL, Gatla S, Wizov SS, Chia T, Spaeth G, Lai S. Structural changes in glaucoma: A volumetric MRI study. Association for Research in Vision and Ophthalmology, 730/A396May 2012.
- [Result] Williams AL, Lackey J, Gatla S, Wizov SS, Sergott R, Chia T, Lai S, Spaeth GL. Correlation of brain volumes and function deficits in glaucoma. 148th Annual AOS Meeting, Charleston, SC 2012.
- [Result] Williams AL. Correlation of brain volumes and patient-reported visual disability in glaucoma. AGS Annual Meeting, San Francisco, March 1, 2012
- [Result] Williams AL, Lackey J, Wizov S, Gatla S, Sergott R, Chia T, Lai S, Spaeth GL. Correlation of brain volumes and functional deficits in glaucoma. Association of Research in Vision and Ophthalmology, 5624 May 10, 2012.
- [Result] Spaeth Gl, Williams AL, Lackey J, Gatla S, Wizov SS, Sergot R, Chia T, Lai S. Glaucoma and the whole patient. AAO 2012 Joint Meeting, Chicago Nov 12, 2012.
- [Result] Williams AL, Lackey J, Wizov SS, Chia TM, Gatla S, Moster ML, Sergott R, Spaeth GL, Lai S. Evidence for widespread structural brain changes in glaucoma: a preliminary voxel-based MRI study. Invest Ophthalmol Vis Sci. 2013 Aug 28;54(8):5880-7. doi: 10.1167/iovs.13-11776. PMID 23838767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 glaucoma patients were enrolled in this study. However, 7 age, gender and ethnic matched controls were not found for study comparisons. Therefore, only the 15 glaucoma patients who best matched the controls were included in the published analysis.
Groups:
- Glaucoma Patients: Patients were outliers from two previous studies: Assessment of Ability Related to Vision (AARV) or Assessment of Disability Related to Vision (ADREV).
- Control Patients: Age, gender and race matched (to the glaucoma patients) group of healthy individuals with no ocular diseases.
Period: Overall Study
Arm/Group | Glaucoma Patients | Control Patients
Started | 22 | 15
Completed | 15 (Matched controls not found for comparisons. Only best matched glaucoma patients were included.) | 15
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Population: All participants completed mini mental status examination with score of 25 or greater then received high resolution 3D T1 weighted magnetic resonance imaging. Seven of the glaucoma patients did not have a control for comparison.
Groups:
- Glaucoma Patients: Patients who were outliers from the AARV or ADREV Studies.
- Control Patients: Age, gender and race matched group of healthy individuals with no ocular diseases.
- Total: Total of all reporting groups
Arm/Group | Glaucoma Patients | Control Patients | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (11.2) | 65.6 (11.3) | 65.85 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Absolute Brain Volume (Size)
Description: Absolute volume (size) of inferior occipital gyrus L (a location in the brain structure) is measured in cubic millimeters (mm3).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm3)
Arm/Group | Glaucoma Patients | Control Patients
Number analyzed (Participants) | 15 | 15
cubic millimeters (mm3) | 3067 (903) | 2302 (357)

2. Secondary Outcome: Relative Volumes
Description: Relative volume is calculated by dividing the absolute volume of inferior occipital gyrus L (a location in the brain structure) by that individual's total brain volume.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: cubic millimeters (mm3)
Arm/Group | Glaucoma Patients | Control Patients
Number analyzed (Participants) | 15 | 15
cubic millimeters (mm3) | 0.0037 (0.001) | 0.0029 (0.001)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Glaucoma Patients | Control Patients
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/15
Other Adverse Events (participants affected / at risk) | 0/22 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No